CLINICAL TRIAL: NCT07101198
Title: Evaluation of the Effectiveness of Ultrasound-Guided Bilateral Erector Spinae Plane Block on Postoperative Pain and Bleeding in Major Spinal Surgery
Brief Title: Ultrasound-Guided Erector Spinae Plane Block in Major Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Funda Atar, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-676
Record Dates: First submitted 2025-07-25; First posted 2025-08-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Perioperative Bleeding; Opioid Consumption; Erector Spinae Plane Block; Spinal Stabilization
Keywords: Spine Surgery; Regional Anesthesia; Blood Loss; Erector Spinae Plane Block
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either ultrasound-guided Erector Spinae Plane Block or no block prior to lumbar spinal stabilization surgery.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded to group assignments. An anesthesiologist not involved in postoperative data collection will perform the Erector Spinae Plane Block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae Plane Block Group (Experimental): Participants in this group received an ultrasound-guided Erector Spinae Plane Block preoperatively as part of multimodal analgesia.
  Interventions: Procedure: Ultrasound-guided erector spinae plane block
- Control Group (No Intervention): Participants in this group did not receive a preoperative regional anesthesia block. Standard postoperative analgesic protocols were used.

INTERVENTIONS:
Procedure: Ultrasound-guided erector spinae plane block — Patients in this group will receive an ultrasound-guided erector spinae plane block 30 minutes before surgery. A total volume of bupivacaine will be injected bilaterally into the fascial plane between the erector spinae muscle and the transverse process. All patients will also receive standard postoperative analgesia.
  Arms: Erector Spinae Plane Block Group

SUMMARY:
This study aims to evaluate the effects of ultrasound-guided bilateral erector spinae plane block on intraoperative pain control and bleeding in patients undergoing major spinal surgery. Participants will be randomly assigned to two groups: one group will receive the Erector Spinae Plane block, while the other group will receive standard pain management. Primary outcomes include postoperative pain levels and intraoperative blood loss. This study seeks to determine whether the Erector Spinae Plane Block technique positively contributes to patient recovery and reduces bleeding complications.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effectiveness of ultrasound-guided bilateral Erector Spinae Plane Block on intraoperative opioid consumption and bleeding in patients undergoing spinal surgery. Eligible adult patients will be enrolled after obtaining informed consent.

Participants will be randomly assigned to two groups: the intervention group will receive bilateral Erector Spinae Plane Block under ultrasound guidance before surgery, while the control group will receive standard pain management without the block. The Erector Spinae Plane Block will be performed using a standard dose of bupivacaine.

The primary outcome measure is the amount of intraoperative bleeding. Secondary outcomes include opioid consumption and incidence of complications.

This study aims to provide evidence on the efficacy of the Erector Spinae Plane Block technique in improving postoperative recovery and reducing bleeding complications in major spinal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older

Scheduled for elective spinal stabilization surgery

American Society of Anesthesiologists (ASA) physical status I-III

Provided written informed consent

Exclusion Criteria: Coagulopathy or current anticoagulant therapy

Anatomical barrier or infection at the Erector Spinae Plane Block site

Known allergy to local anesthetics or opioids

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-07-24 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Intraoperative estimated blood loss | During surgery
  Intraoperative estimated blood loss (milliliters) Total amount of blood lost during surgery will be measured in milliliters. [Time Frame: During surgery]

SECONDARY OUTCOMES:
Total intraoperative remifentanil consumption | During surgery
  The total dose of remifentanil administered intraoperatively (in micrograms) will be recorded by the anesthesia team.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Atar, MD, Principal Investigator — Ankara Etlik City Hospital; Derya Özkan, prof, Study Director — Ankara Etlik City Hospital
Locations (1):
- Etlik city hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No